CLINICAL TRIAL: NCT05155436
Title: Prevalence and Incidence of Dyskalemia in Hypertensive Patients Initiating a Fixed Dose Combination Pill of Telmisartan and Amlodipine
Brief Title: Occurrence of Dyskalemia With Treatment for Hypertension
Acronym: OK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Heart Foundation of Bangladesh (Other)
Collaborators: National Heart Foundation Hospital and Research Institute of Bangladesh (Unknown); Johns Hopkins University (Other); Resolve to Save Lives (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210921/4
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Hypertension; Potassium Imbalance
Keywords: Hyperkalemia; Hypertension; Hypokalemia
MeSH Terms: conditions — Hypertension; Hyperkalemia; Hypokalemia | interventions — Telmisartan; Amlodipine

STUDY DESIGN:
Intervention Model Description: The people residing in Mirpur at Dhaka city have been included in this study with matching the inclusion criteria which are as follows: Age ≥40 years for men and ≥ 50 years for women who had menopause for 1 year; Systolic blood pressure (SBP) ≥140 mmHg and/or diastolic blood pressure (DBP) ≥90 mmHg (average across two visits as detailed in 'Measurements' section below); Adults not currently (in the past month) taking BP medications
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fixed-Dose Combination pill of Telmisartan and Amlodipine (Experimental): Fixed-Dose Combination pill of Telmisartan 40 mg and Amlodipine 5 mg, once daily for 3 months
  Interventions: Drug: Fixed Dose Combination pill of Telmisartan 40mg and Amlodipine 5 mg

INTERVENTIONS:
Drug: Fixed Dose Combination pill of Telmisartan 40mg and Amlodipine 5 mg — Participants without prevalent hyperkalemia will receive the fixed-dose combination pill of Telmisartan and Amlodipine, once daily for 3 months.

SUMMARY:
Hypertension is a major public health issue associated with significant morbidities and mortality. Fixed-dose combination (FDC) pills, combining 2 or more classes of antihypertensive medications have considerable appeal because these drugs may reduce blood pressure more effectively and efficiently compared to monotherapy. However, because FDC medication causes 'dyskalemia', the occurrence of either hypo- or hyper-kalemia, which requires laboratory testing, implementing FDC is hampered in some low- and middle-income countries where laboratory testing is limited. This study will be conducted in the area of Mirpur in Dhaka, Bangladesh, to 1) estimate the prevalence of dyskalemia in hypertensive patients who are candidates for pharmacotherapy; and 2) of those patients initiating a FDC combining telmisartan 40 mg/amlodipine 5 mg, estimate the incidence of dyskalemia at two months later. Telmisartan is a widely prescribed drug approved by the Directorate General of Drug Administration (DGDA). If the prevalence and incidence of dyskalemia is low, as anticipated, this study results will provide evidence that routine laboratory testing might not be necessary. It is to be mentioned that Telmisartan is not a new drug and it is a widely prescribed drug approved by the Directorate General of Drug Administration (DGDA), Bangladesh

DETAILED DESCRIPTION:
Hypertension affects an estimated 1.04 billion people in low- and middle-income countries, with an estimated increase in prevalence of 7.7% between 2000 and 2010.1 Hypertension treatment and control may lower the risk of cardiovascular disease and mortality by 20-40%.2 However, less than 10% of individuals with hypertension are under control in low- and middle-income countries, contributing to substantial morbidity and mortality.1 The low prevalence of controlled hypertension may be partly because the vast majority (85.5%) of hypertensive individuals in low- and middle-income countries receive a monotherapy,3 although two or more medications are often needed to achieve a target blood pressure.4 Fixed dose combination (FDC) pills, combining 2 or more classes of antihypertensive medications have considerable appeal because these may reduce blood pressure (BP) more effectively and efficiently compared to monotherapy by blocking two pathways contributing to hypertension.5 Systematic reviews and meta-analyses have shown that FDC pills decreased the risk of non-compliance by 26% compared with free-drug component regimen, while keeping the same rate of reduction in the risk of cardiovascular events.6,7 However, many effective FDC antihypertensive medications include either or both thiazide/thiazide-like diuretic and a renin-angiotensin system inhibitor (RASI) and use of these medications alone, or in combination, generally require laboratory tests to monitor serum potassium. The principal metabolic concern is a risk of incident 'dyskalemia', the occurrence of either hypo- or hyper-kalemia: diuretic-induced hypokalemia and RASI-induced hyperkalemia. Practice guidelines commonly recommend laboratory testing prior to initiation of these drugs, alone or as part of FDC, and periodic monitoring during medication treatment, but guidelines are extremely inconsistent8,9 and are not routinely implemented.10,11 The requirement for laboratory testing is an impediment to implementing FDC in low- and middle-income countries. Therefore, this study will quantify the risk (i.e., prevalence and incidence) of dyskalemia in the context of FDC medication as initial therapy. The study is designed to implement a promising FDC antihypertensive medication of angiotensin receptor blocker (ARB, telmisartan) and calcium channel blocker (CCB, amlodipine) in Bangladesh clinics in collaboration among the National Heart Foundation of Bangladesh, Resolve to Save Lives, and Johns Hopkins University.

Objectives:

* To estimate the prevalence of dyskalemia in hypertensive patients who are candidates for pharmacotherapy.
* Of those patients initiating antihypertensive medication, estimate the incidence of dyskalemia at two months after initiating an FDC combining telmisartan 40 mg/amlodipine 5 mg.

Study Design:

This study will be pre-post study design. This design is chosen because the incidence of dyskalemia is reasonably considered attributable to the initiation of FDC medication, given the short follow-up period (i.e., the only change is the initiation of FDC medication in the exposure status, and it is unlikely that other significant changes in medical and health conditions occur and subsequently impact the incidence of dyskalemia). Because each individual can serve as both control and treatment (i.e., the prevalence of dyskalemia will serve as the control), the pre-post design will be efficient to address this research question while reserving the scientific rigor, compared to randomized control trials, which would require a much larger sample size.

Participants: The study will enroll adults (aged ≥40 years for men and ≥50 years for women) with hypertension in Bangladesh who are eligible for the initiation of antihypertensive medication. The age criteria are chosen because middle-aged to older adults bear the major burden of dyskalemia. Due to the concern of teratogenicity of angiotensin receptor blockers, this study will not include women aged <50 years in the study. This cut-off was selected based on the general consideration of reproductive age (e.g., 15-44 years in reports by the United States Centers for Disease Control and Prevention). this study also will not recruit individuals who are unable to provide informed consent (e.g., children).

Intervention:

Participants without prevalent hyperkalemia will receive the FDC telmisartan 40 mg/amlodipine 5 mg combination pill (1 pill a day). The cost for FDC per tablet is 12 to 15 cents, but study participants will receive the study medication free of charge for three months. A combination of telmisartan and amlodipine was selected according to the World Health Organization (WHO) Model List of Essential Medicine.17 Of note, two-drug FDC pills of ARB and CCB for hypertension were recently added to the WHO Model List of Essential Medicine to improve global availability and affordability, following an application from the Resolve To Save Lives.6

Measurements:

There will be four (04) study visits for the study: screening visit, eligibility visit, FDC initiation visit, and follow-up visit.

Adherence and retention strategy:

General strategy: The study is designed to promote high adherence and retention, e.g., few visits, low data collection burden, and brief study duration. During implementation, this study will actively promote adherence at the in-person visits and telephone calls. The first call will happen approximately 1 week after the FDC initiation visit. The investigators will check in on participants to see if the participants have any issues or concerns after taking the medication. The second call will happen just before the follow-up visit. The main purpose of this second call is to encourage participants to return to the clinic for follow-up visits. In addition to active phone-calls to participants, there will be setting up of a hotline so that participants can contact the clinic when the participants have questions or concerns.

Safety monitoring strategy:

The principal risks of the study are symptoms and adverse effects related to the FDC, primarily hypotension. When adverse events are suspected (e.g., dizziness), participants will be advised to call us on the hotline. Depending on the nature of the symptom, participants will be asked to visit the clinic. Study physicians will evaluate the participant and may adjust the medication if needed (e.g., switch to amlodipine monotherapy or stop medication). In such scenarios, lab tests will be conducted at the timing of medication adjustment/discontinuation and will include these participants in the primary analysis (regardless of the duration of follow-up). Serious adverse events, defined by the United States Food and Drug Administration,19 will be collected and reported to the data safety and monitoring board.

Potential risks and strategies to mitigate the risks:

This study anticipates minimal psychological or physical risks to participants. The major anticipated risks and strategies to mitigate the risks are Loss of confidentiality, Blood pressure measurement, Blood draw, Blood pressure medication.

Sample size calculation:

In order to detect a dyskalemia incidence of 2.5% or higher, the study will need to enroll 1,290 participants who are free of dyskalemia at screening and who complete a follow-up visit, assuming a type I error probability of 0.05 (two-sided) and 80% power.). For this calculation, the threshold of 2.5% corresponds to the 'tolerable limit', which is the level that would be deemed unacceptable based on available literature and assessment of the study's clinician investigators10,11 its estimated that if the observed incidence of dyskalemia is 1.5%, then the actual incidence will not exceed 2.5%.

Analysis plan:

The analysis will be performed jointly between Bangladesh and Hopkins team. Descriptive statistics will be presented as mean (SD) for continuous variables and numbers (percentage) for categorical variables. this study will use histograms to describe the distribution of potassium levels prior to and after the initiation of FDC medication. The prevalence and incidence of dyskalemia, and other binary outcomes of interest will be estimated using Poisson regression models

Data management:

Data entry process At screening sites, paper-based questionnaire forms will be filled by participants. Then, project staff (interviewers) will enter the data into Redcap. At clinics, the clinic nurses will conduct an interview and record the response on a mobile computing device into Redcap. All data will be saved in the server of NHFB.

Data management The Research Officer of the study clinic will be the designated person for data management. Study personnel and the principal investigators will be responsible for monitoring and evaluating the completeness of data. Suspected missing data and discrepancies will be reported to the study site, and necessary corrections will be requested.

Facilities

National Heart Foundation Hospital & Research Institute, Screening room, Hypertension Clinic, Pathological Laboratory with all apparatus and chemical reagents required for blood and urine test. Additional Facilities Required: No additional facilities are required.

Utilization of results

This project will provide valuable information related to the need, if any, for laboratory testing prior to and during the treatment of patients with hypertension who are candidates for medication treatment. Findings from this study could change the approach to managing hypertension and ultimately lead to improved hypertension control which subsequently reduces the risk of cardiovascular disease in this population. In addition, results deriving from this project will also be shared in several ways. the investigators will publish the study results in peer-reviewed journals. In addition, findings including preliminary data will be presented at national conferences.

Ethical implications

The study will be conducted as part of usual care for hypertension, and participants will benefit from treating hypertension through the use of FDC medication. Additionally, the study findings, the incidence of dyskalemia after initiating FDC medication, could ultimately contribute to the significant public health benefits. Specifically, if the prevalence and incidence of dyskalemia is low, as anticipated, this study results will provide evidence that routine laboratory testing might not be necessary. Given that this study poses minimal risk and inconvenience to participants, this study anticipates the potential risks are outweighed by the benefits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40 years for men and ≥ 50 years for women who had menopause for 1 year
* Systolic blood pressure (SBP) ≥140 mmHg and/or diastolic blood pressure (DBP) ≥90 mmHg (average across two visits as detailed in 'Measurements' section below)
* Adults not currently (in the past month) taking BP medications

Exclusion Criteria:

* SBP of ≥180 mmHg, DBP of ≥120 mmHg
* Creatinine clearance (Cockcroft-Gault Equation) <30 ml/min
* Serum potassium >5 or <3 mmol/L
* History of intolerance or allergy to ACEI, ARB, or calcium channel blockers
* Women who are currently pregnant, or planning to become pregnant
* Women who are currently breastfeeding
* Other serious conditions (e.g., those with heart failure treated with medication, COPD patients using Salbutamol etc)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1090 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Prevalent dyskalemia at baseline in patients eligible for antihypertensive medications. | 2 months from administration of intervention
  to find out the prevalence of dyskalemia at baseline in patients eligible for antihypertensive medications.
Incident dyskalemia after 2 months of therapy (dyskalemia defined as a follow-up serum potassium < 3.0 or > 5.5 mmol/L | 2 months from administration of intervention
  to estimate the number of patients with dyskalemia after administration of FDC for 2 months.

SECONDARY OUTCOMES:
Hyperkalemia alone | 2 months from administration of intervention
  to estimate the number of patients with high potassium level (>5 mmol/l) after administration of FDC for 2 months.
Hypokalemia alone | 2 months from administration of intervention
  to estimate the number of patients with low potassium (<3 mmol/l) after administration of FDC for 2 months.
Blood pressure change | 2 months from administration of intervention
  to estimate the number of patients with any changes in blood pressure after administration of FDC for 2 months.
Adherence | 2 months from administration of intervention
  to estimate the number of patients took medicine regularly as instructed.

CONTACTS AND LOCATIONS:
Overall Officials: Fazilatunnesa Malik, MBBS, FCPS, Principal Investigator — National Heart Foundation, Bangladesh
Locations (1):
- National Heart Foundation of Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abernethy DR. Pharmacokinetics and pharmacodynamics of amlodipine. Cardiology. 1992;80 Suppl 1:31-6. doi: 10.1159/000175050. PMID 1534713
- [Background] Bandak G, Sang Y, Gasparini A, Chang AR, Ballew SH, Evans M, Arnlov J, Lund LH, Inker LA, Coresh J, Carrero JJ, Grams ME. Hyperkalemia After Initiating Renin-Angiotensin System Blockade: The Stockholm Creatinine Measurements (SCREAM) Project. J Am Heart Assoc. 2017 Jul 19;6(7):e005428. doi: 10.1161/JAHA.116.005428. PMID 28724651
- [Background] Bangalore S, Kamalakkannan G, Parkar S, Messerli FH. Fixed-dose combinations improve medication compliance: a meta-analysis. Am J Med. 2007 Aug;120(8):713-9. doi: 10.1016/j.amjmed.2006.08.033. PMID 17679131
- [Background] Betts KA, Woolley JM, Mu F, McDonald E, Tang W, Wu EQ. The prevalence of hyperkalemia in the United States. Curr Med Res Opin. 2018 Jun;34(6):971-978. doi: 10.1080/03007995.2018.1433141. Epub 2018 Feb 21. PMID 29368958
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. National Heart, Lung, and Blood Institute; National High Blood Pressure Education Program Coordinating Committee. Seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Hypertension. 2003 Dec;42(6):1206-52. doi: 10.1161/01.HYP.0000107251.49515.c2. Epub 2003 Dec 1. PMID 14656957
- [Background] Chow CK, Teo KK, Rangarajan S, Islam S, Gupta R, Avezum A, Bahonar A, Chifamba J, Dagenais G, Diaz R, Kazmi K, Lanas F, Wei L, Lopez-Jaramillo P, Fanghong L, Ismail NH, Puoane T, Rosengren A, Szuba A, Temizhan A, Wielgosz A, Yusuf R, Yusufali A, McKee M, Liu L, Mony P, Yusuf S; PURE (Prospective Urban Rural Epidemiology) Study investigators. Prevalence, awareness, treatment, and control of hypertension in rural and urban communities in high-, middle-, and low-income countries. JAMA. 2013 Sep 4;310(9):959-68. doi: 10.1001/jama.2013.184182. PMID 24002282
- [Background] Chowdhury MZI, Rahman M, Akter T, Akhter T, Ahmed A, Shovon MA, Farhana Z, Chowdhury N, Turin TC. Hypertension prevalence and its trend in Bangladesh: evidence from a systematic review and meta-analysis. Clin Hypertens. 2020 Jun 1;26:10. doi: 10.1186/s40885-020-00143-1. eCollection 2020. PMID 32514373
- [Background] Ettehad D, Emdin CA, Kiran A, Anderson SG, Callender T, Emberson J, Chalmers J, Rodgers A, Rahimi K. Blood pressure lowering for prevention of cardiovascular disease and death: a systematic review and meta-analysis. Lancet. 2016 Mar 5;387(10022):957-967. doi: 10.1016/S0140-6736(15)01225-8. Epub 2015 Dec 24. PMID 26724178
- [Background] Guerrero-Garcia C, Rubio-Guerra AF. Combination therapy in the treatment of hypertension. Drugs Context. 2018 Jun 6;7:212531. doi: 10.7573/dic.212531. eCollection 2018. PMID 29899755
- [Background] Kishore SP, Salam A, Rodgers A, Jaffe MG, Frieden T. Fixed-dose combinations for hypertension. Lancet. 2018 Sep 8;392(10150):819-820. doi: 10.1016/S0140-6736(18)31814-2. No abstract available. PMID 30215377
- [Background] Lewington S, Clarke R, Qizilbash N, Peto R, Collins R; Prospective Studies Collaboration. Age-specific relevance of usual blood pressure to vascular mortality: a meta-analysis of individual data for one million adults in 61 prospective studies. Lancet. 2002 Dec 14;360(9349):1903-13. doi: 10.1016/s0140-6736(02)11911-8. PMID 12493255
- [Background] Littlejohn TW 3rd, Majul CR, Olvera R, Seeber M, Kobe M, Guthrie R, Oigman W; Study Investigators. Results of treatment with telmisartan-amlodipine in hypertensive patients. J Clin Hypertens (Greenwich). 2009 Apr;11(4):207-13. doi: 10.1111/j.1751-7176.2009.00098.x. PMID 19614805
- [Background] Mills KT, Bundy JD, Kelly TN, Reed JE, Kearney PM, Reynolds K, Chen J, He J. Global Disparities of Hypertension Prevalence and Control: A Systematic Analysis of Population-Based Studies From 90 Countries. Circulation. 2016 Aug 9;134(6):441-50. doi: 10.1161/CIRCULATIONAHA.115.018912. PMID 27502908
- [Background] Osmundson SS, Gould JB, Butwick AJ, Yeaton-Massey A, El-Sayed YY. Labor outcome at extremely advanced maternal age. Am J Obstet Gynecol. 2016 Mar;214(3):362.e1-7. doi: 10.1016/j.ajog.2015.09.103. Epub 2015 Nov 18. PMID 26454124
- [Background] Parikh RV, Nash DM, Brimble KS, Markle-Reid M, Tan TC, McArthur E, Khoshniat-Rad F, Sood MM, Zheng S, Pravoverov L, Nesrallah GE, Garg AX, Go AS. Kidney Function and Potassium Monitoring After Initiation of Renin-Angiotensin-Aldosterone System Blockade Therapy and Outcomes in 2 North American Populations. Circ Cardiovasc Qual Outcomes. 2020 Sep;13(9):e006415. doi: 10.1161/CIRCOUTCOMES.119.006415. Epub 2020 Sep 2. PMID 32873054
- [Background] Unger T, Borghi C, Charchar F, Khan NA, Poulter NR, Prabhakaran D, Ramirez A, Schlaich M, Stergiou GS, Tomaszewski M, Wainford RD, Williams B, Schutte AE. 2020 International Society of Hypertension global hypertension practice guidelines. J Hypertens. 2020 Jun;38(6):982-1004. doi: 10.1097/HJH.0000000000002453. No abstract available. PMID 32371787
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):1269-1324. doi: 10.1161/HYP.0000000000000066. Epub 2017 Nov 13. No abstract available. PMID 29133354